CLINICAL TRIAL: NCT02471573
Title: The Effectiveness of a Freeze All Protocol Versus Fresh Embryo Transfer in Women Undergoing In-vitro Fertilization (IVF) - Intracytoplasmic Sperm Injection (ICSI)
Brief Title: Freeze All Protocol Versus Fresh Embryo Transfer in Women Undergoing In-vitro Fertilization (IVF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam National University (Other)
Collaborators: Mỹ Đức Hospital (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Doctor, Vietnam National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCKH/CGRH_ 03_2015
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Infertility
Keywords: IVF; Freeze-all; frozen embryo transfer; fresh transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Freeze-all protocol (Active Comparator): Embryos are selected for cryopreservation using vitrification technique. Two vitrified embryos will be warmed and transferred in subsequent cycle.
  Interventions: Procedure: Freeze-all protocol
- Fresh transfer protocol (Active Comparator): Two embryos are selected and transferred fresh in the same cycle.
  Interventions: Procedure: Fresh transfer protocol

INTERVENTIONS:
Procedure: Freeze-all protocol — Embryos are selected for cryopreservation using vitrification technique. Two vitrified embryos will be warmed and transferred in subsequent cycle.
  Arms: Freeze-all protocol
Procedure: Fresh transfer protocol — Two embryos are selected and transferred fresh in the same cycle.
  Arms: Fresh transfer protocol

SUMMARY:
To compare the effectiveness of freeze-all and subsequent frozen embryo transfer (freeze all protocol) with fresh embryo transfer (fresh ET).

DETAILED DESCRIPTION:
All patients undergoing in-vitro fertilization (IVF) will be treated with GnRH antagonist protocol. Recombinant Follicle-stimulating hormone (FSH) will be given on day 2 or day 3 of menstrual cycle for 5 days. The starting dose is individualized for each patient based on the following criteria: Anti-Mullerian Hormone (AMH) < 0.7 ng/ml, dose 300 IU/day, AMH 0.7 -2.1 ng/ml, dose 225 IU/day, AMH > 2.1 ng/ml, dose 150 IU/day. After that, investigators can titrate the dose based on their clinical judgment. Follicular development will be monitored by ultrasound scanning and measurement of estradiol, progesterone starting on day 5 of stimulation. Scanning and hormonal measurement will be repeated every 2 to 3 days, depending on the size of follicles. Antagonist is routinely used on day 5 until the day of Human chorionic gonadotropin (hCG). Criteria for recombinant hCG (6,500 IU) administration is the presence of at least three leading follicles of 17 mm. Oocyte retrieval is performed 36 hours after recombinant hCG administration.

We will measure progesterone levels during stimulation on the day 5 and day 7, as well as on the day of oocyte triggering.

Insemination will be performed by using intracytoplasmic sperm injection, 3 - 4 hours after oocyte retrieval. Only matured oocytes are inseminated. Fertilization are performed under inverted microscope at period of 16-18 hours after insemination.

On day 3, endometrium thickness will be measured and embryo evaluation will be performed at fixed time point 68±1 hours after fertilization, using Istanbul consensus. After grading embryo, eligible patients will be invited to participate in the study. Written consent will be obtained from each patient for participation into the study. Patients will be randomized into 2 groups fresh embryo transfer and freeze-all. Randomization will be done by third party via telephone, using a computer-generated random list, with block size of 2, 4, 8.

Study Procedures

Freeze all group

All grade 1 and grade 2 embryos were cryopreserved using vitrification method. In the next cycle, endometrium will be prepared by using estradiol orally, starting from day 2-3 of menstrual cycle. When endometrium thickness reaches 8mm or more, patients start to use progesterone vaginally. Embryo transfer is performed 3 days after using progesterone. On the day of embryo transfer, maximum two embryos will be thawed. Two hours after thawing, surviving embryos will be transferred into the uterus under ultrasound guidance. Luteal-phase support is done with estradiol 8mg/day and vaginal progesterone 800mg/day until 7th week of gestation.

Fresh ET group

In fresh ET group, maximum 2 embryos will be transferred into the uterus under ultrasound guidance. The remain grade 1 and 2 embryos will be frozen. Luteal phase support is done with estradiol 8mg/day and vaginal progesterone 800mg/day until 7th week of gestation.

In both of groups, serum hCG was measured 2 weeks after embryo transferred, and if positive, an ultrasound scan of the uterus was performed at gestational weeks 7 and 12.

METHODS

SAMPLE SIZE CALCULATION

At IVFMD, the current ongoing pregnancy rate (with 2 embryos transferred) is 30%. To show an improvement in the freeze-all group of 10% (from 30% to 40%), it was calculated that 712 couples (356 in each group) would be needed (power 0.80, alpha-error 5%, two-sided test). To account for an estimated loss to follow-up rate of 10%, the number of patients needed was defined as 780 (390 patients per group).

STUDY ENDPOINTS

Primary endpoint

Ongoing pregnancy (OP). Ongoing pregnancy is explained as a pregnancy with positive heart beat beyond 12 weeks of gestation (twins is count as a single pregnancy).

Secondary endpoints

* Implantation rate: defined as the number of gestational sacs per number of embryos transferred.
* Clinical pregnancy: defined as the presence of a gestational sac seen by transvaginal sonography 7 weeks after embryo replacement.
* Multiple pregnancy rate. defined as a pregnancy with two or more fetal heart beats by transvaginal sonography at 7 weeks of gestation.
* Vanishing twins: defined as a pregnancy with tow or more gestational sacs or positive heart beats at 7 weeks of gestation, but only one at 12 weeks' gestation.

Treatment complications

* Ovarian hyperstimulation syndrome (OHSS): classified as moderate or severe by RCOG guidelines [Green-top Guideline No. 5, 2006].
* Miscarriage: defined as the complete loss of a clinical pregnancy prior to 24 weeks' gestation.
* Ectopic pregnancy: defined as the ectopic nidation of a pregnancy, confirmed by sonography or laparoscopy.

Obstetric outcomes

* Live birth rate, defined as the birth of a newborn, irrespective of the duration of gestation, that exhibits any sign of life, such as respiration, heart-beat, umbilical pulsation or movement of voluntary muscles.
* Gestational age at delivery.
* Birth weight.
* Congenital malformations.
* Macrosomia (birth weight >90th percentile)
* Small for gestational age (birth weight <10th percentile)
* NICU admittance
* Perinatal mortality: defined as the death of a fetus or infant from 24 weeks of gestation to the end of the neonatal period of 4 weeks after birth.

Pregnancy complications

* Pregnancy-associated hypertension: defined as a diagnosis of pregnancy-induced hypertension made after the 20th week of gestation, excluding intraoperative blood pressures and intrapartum systolic pressures, with systolic blood pressure of ≥140 mmHg or diastolic pressure of ≥90 mmHg on two occasions 2 hours apart, or a severely elevated single blood pressure measurement that led to treatment with an antihypertensive medication.
* Preeclampsia: defined as any type of hypertension combined with proteinuria (total protein excretion of 300 mg or other organ involvement [such as renal insufficiency, liver involvement, neurological or hematological complications, uteroplacental dysfunction, or fetal growth restriction]) according to the International Society of Studies in Hypertension in Pregnancy.
* HELLP syndrome: defined as elevated liver enzyme levels (aspartate aminotransferase ≥100 U/L), thrombocytopenia (platelet count <100,000/mm3), elevated serum creatinine level (≥1.5 mg/dL [132.6 μmol/L]) and/or hemolysis (hemoglobin <10 g/dL).
* Prematurity: defined as iatrogenic preterm birth at <32 weeks' gestation, spontaneous preterm birth at <32 weeks' gestation; iatrogenic preterm birth at <37 weeks gestation; spontaneous preterm birth at <37 weeks' gestation
* Antepartum hemorrhage: defined as bleeding from the genital tract in the second half of pregnancy.
* Gestational diabetes mellitus: diagnosed using a 75g oral glucose tolerance test (Fasting: 92 mg/dL [5.1 mmol/L]; 2 h: 153 mg/dL [8.5 mmol/L]) [American Diabetes Association 2013].

Labor

Induction of labor

* Cesarean section

  * Elective
  * Suspected fetal distress
  * Non-progressive labor
* Vaginal instrumental delivery

  * Suspected fetal distress
  * Non-progressive labor
* Peripartum increased blood loss (≥1000 mL)

SUBJECT INFORMED CONSENT A review of patient information should be done prior to enrolment to determine preliminary eligibility according to patient inclusion and exclusion criteria. When a patient signs an informed consent she is considered to be enrolled in the study.

WITHDRAWAL OF INDIVIDUAL PATIENTS Patients can leave the study at any time for any reason if they wish to do so without any consequences for their treatment. The investigator can decide to withdraw a subject from the study or urgent medical reasons.

STATISTICAL EVALUATION

Event rates will be calculated for dichotomous endpoints. These will be compared by calculating relative risk and 95% confidence interval values. Between-group differences in non-continuous variables will be assessed using the Fisher exact test. Continuous variables will be reported as mean values ± standard deviation (SD) or as percentages. Between-group differences in continuous variables will be assessed with the Student's t-test.

In a secondary analysis we will assess whether the biomarkers progesterone at triggering day and endometrial thickness on day 3 after oocyte pick up can be used to identify patients in whom the freeze all strategy is particularly effective. To do so, we will look for interaction between progesterone or endometrial thickness and treatment effect.

A p-value <0.05 is defined as indicating a statistically significant difference. The analysis will be done with R statistical package (R version 3.3.1).

INTERIM ANALYSIS

Interim analysis will be performed after recruitment of the first 400 patients. An independent Data Safety Monitoring Committee (DSMC) will evaluate the data. A specific stopping rule will not be formulated, but continuation of the study will depend on the advice of the DSMC.

SAFETY REPORTING

The investigator will inform the subjects and the reviewing accredited medical research ethics committee; if anything occurs, on the basis of which it appears that the disadvantages of participation may be significantly greater than was foreseen in the research proposal. The investigator will take care that all subjects are kept informed.

ADVERSE AND SERIOUS ADVERSE EVENTS All observed or volunteered adverse events, regardless of treatment group or suspected causal relationship to intervention, will be recorded. Adverse events are defined as any undesirable experience occurring to a subject during a clinical trial, whether or not considered related to the intervention. All adverse events reported spontaneously by the subject or observed by the investigator or his staffs will be recorded.

A serious adverse event is any untoward medical occurrence or effect that at any dose results in death;

* is life threatening (at the time of the event);
* requires hospitalisation or prolongation of existing inpatients' hospitalisation;
* results in persistent or significant disability or incapacity;
* is a congenital anomaly or birth defect;
* is a new event of the trial likely to affect the safety of the subjects, such as an unexpected outcome of an adverse reaction.

ETHICAL CONSIDERATIONS

RECRUITMENT AND CONSENT The subject should be given the time to read and understand the statement herself before signing her consent and dating the document. The subject should receive a copy of the written statement once signed.

PRIVACY ASPECTS Participating subjects will be registered by a 5-digit number. This personal code will be on all forms retrieved from participants.

BENEFITS AND RISKS ASSESSMENT, GROUP RELATEDNESS There is insufficient evidence for a rational policy in between the 2 strategies, freeze all or fresh ET. The potential benefits of freeze all are higher pregnancy rate, with a lower incidence of ovarian hyperstimulation syndrome (OHSS) and/or ectopic pregnancy. The potential harm would be time-consuming.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing In-vitro fertilization (IVF) treatment
* Number of previous failed embryo transfers ≤ 2
* Permanent living in Viet Nam
* Ovarian hyperstimulation with Gonadotropin releasing hormone (GnRH) antagonist protocol
* Eligible for embryo transfer (ET) on day 3
* Having at least one top-quality embryo on day 3.
* Number of embryos transferred ≤ 2
* Willing to participate in the study
* Not to participate in another IVF study at the same time

Exclusion Criteria:

* women with polycystic ovary syndrome
* In vitro maturation (IVM) cycles
* Oocyte donation cycles
* Using GnRH agonist for triggering

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 782 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2016-04-10 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy | 12 weeks of gestation
  Ongoing pregnancy is defined as a pregnancy with at least one positive heart beat beyond 12 weeks of gestation.

SECONDARY OUTCOMES:
Clinical pregnancy | 5 weeks after embryo placement
  Clinical pregnancy is explained as the presence of a gestational sac seen by transvaginal sonography.
Implantation rate | 3 weeks after embryo transferred
  Implantation rate is explained as as the number of gestational sacs per number of embryos transferred.
Multiple pregnancy rate | 5 weeks after embryo placement
  Multiple pregnancy is explained as two or more gestational sacs or positive heart beats by transvaginal sonography.
Live birth | at the time of delivery
  Live birth is defined if a live newborn delivered.

OTHER OUTCOMES:
Ovarian hyperstimulation syndrome (OHSS) | at 10 days after hCG injection and 14 days after embryo transfer
  Symptoms of OHSS
Miscarriage | at 24 weeks of gestation
  complete lost of clinical pregnancy
Ectopic pregnancy | at 12 weeks of gestation
  ectopic nidation of a pregnancy confirmed by sonography or laparoscopy
Live birth | at birth
  birth of a newborn with any sign of life
Gestational age at delivery | at the time of delivery
  gestational age at delivery
Birth weight | at the time of delivery
  Weight of newborn
congenital malformation | at the time of delivery
  congenital malformation of newborn
Macrosomia | at the time of delivery
  Birth weight > 90th percentile
small for gestational age | at the time of delivery
  birth weight < 10th percentile
NICU admittance | 7 days after delivery
  The admittance of the newborn to NICU
Pregnancy-associated hypertension | at 20 weeks of gestation
  systolic blood pressure of ≥140 mmHg or diastolic pressure of ≥90 mmHg on two occasions 2 hours apart, or a severely elevated single blood pressure measurement that led to treatment with an antihypertensive medication.
Preeclampsia | at 20 weeks of gestation
  any type of hypertension combined with proteinuria (total protein excretion of 300 mg or other organ involvement [such as renal insufficiency, liver involvement, neurological or hematological complications, uteroplacental dysfunction, or fetal growth restriction])
HELLP syndrome | at 20 weeks of gestation
  elevated liver enzyme levels (aspartate aminotransferase ≥100 U/L), thrombocytopenia (platelet count <100,000/mm3), elevated serum creatinine level (≥1.5 mg/dL [132.6 μmol/L]) and/or hemolysis (hemoglobin <10 g/dL)
Prematurity | at 32 weeks and 37 weeks of gestation
  Preterm birth
antepartum hemorrhage | in the second half of pregnancy
  bleeding from the genital tract
Gestational diabetes mellitus | at 24 weeks of gestation
  using a 75g oral glucose tolerance test
Mode of deliver | at the time of delivery
  Normal delivery, vaginal instrument delivery or Cesarean section
Permpartum increased blood loss | 24 hours after delivery
  Blood loss more than 1000ml

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Study Chair — Research Center for Genetics and Reproductive Health, School of Medicine, Vietnam National University HCMC
Locations (1):
- My Duc Hospital, IVFMD, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zaat T, Zagers M, Mol F, Goddijn M, van Wely M, Mastenbroek S. Fresh versus frozen embryo transfers in assisted reproduction. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD011184. doi: 10.1002/14651858.CD011184.pub3. PMID 33539543
- [Derived] Vuong LN, Ly TT, Nguyen NA, Nguyen LMT, Le XTH, Le TK, Le KTQ, Le TV, Nguyen MHN, Dang VQ, Norman RJ, Mol BW, Ho TM. Development of children born from freeze-only versus fresh embryo transfer: follow-up of a randomized controlled trial. Fertil Steril. 2020 Sep;114(3):558-566. doi: 10.1016/j.fertnstert.2020.04.041. Epub 2020 Jun 16. PMID 32560970
- [Derived] Vuong LN, Dang VQ, Ho TM, Huynh BG, Ha DT, Pham TD, Nguyen LK, Norman RJ, Mol BW. IVF Transfer of Fresh or Frozen Embryos in Women without Polycystic Ovaries. N Engl J Med. 2018 Jan 11;378(2):137-147. doi: 10.1056/NEJMoa1703768. PMID 29320655